CLINICAL TRIAL: NCT03621293
Title: Long Term Outcome on Brain and Lung of Different Oxygen Strategies in ARDS Patients
Acronym: LTO-BLOXY
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: N/2016/74
Record Dates: First submitted 2018-08-01; First posted 2018-08-08 (Actual); Last update posted 2018-08-08 (Actual); Status verified 2018-08

CONDITIONS: Acute Respiratory Distress Syndrome
Keywords: Long term outcome; Brain; Lung; Oxygen strategies
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Liberal Oxygenation (LO) group (Active Comparator): A modulation of inspired fraction of oxygen will be performed with an objective of PaO2 between 90 to 105 mmHg that will be checked on arterial blood gases (ABG). Between these measurements, SpO2 will be kept more or equal to 96 percent. Alarms will be set at 95 percent for SpO2.
  Intervention: Drug: Modulation of Inspired Fraction of Oxygen (FiO2)
  Interventions: Drug: Modulation of Inspired Fraction of Oxygen (FiO2)
- Conservative Oxygenation (CO) group (Experimental): A modulation of inspired fraction of oxygen will be performed with an objective of PaO2 between 55 to 70 mmHg that will be checked on arterial blood gases. Between these measurements, SpO2 will be kept between 88 and 92 percent. Alarms will be set between 87 and 93 percent for SpO2.
  Intervention: Drug: Modulation of Inspired Fraction of Oxygen (FiO2)
  Interventions: Drug: Modulation of Inspired Fraction of Oxygen (FiO2)

INTERVENTIONS:
Drug: Modulation of Inspired Fraction of Oxygen (FiO2) — In the two groups, if patient is not in the range of arterial oxygen pressure (PaO2), Inspired Fraction of Oxygen (FiO2) will be modified from 5 percent if difference between target is less than 5 mmHg and from 10 percent if difference from target is higher. A new arterial blood gases (ABG) will be performed 30 minutes later to check for the oxygen target range. When ABG are performed, pulsed oxymetry is compared with arterial saturation (SaO2) to adapt survey. Between each ABG, FiO2 is modified from 5 percent to 5 percent each five minutes until reaching good pulsed oxygen saturation (SpO2) target (that can be modified in function of the comparison of arterial oxygen saturation (SaO2 and SpO2 with ABG).
  This management of FiO2 will be done until extubation of the patient.

SUMMARY:
Acute respiratory distress syndrome (ARDS) is a serious disease with high mortality. In patients who survive ARDS, respiratory, neurological and motor sequelae are frequent, negatively impacting on the patient's quality of life, and engendering substantial healthcare costs (rehabilitation, long-term care, delayed return to work). There may also be repercussions on the patient's family and entourage. The severity of ARDS and the burden it represents have underpinned intensive research to identify treatment strategies that could improve mortality. However, it is important to ensure that any improvement in mortality does not come at the price of an excess of sequelae and disability in survivors.

The oxygenation strategy used to treat ARDS may have an impact on mortality in these patients. The CLOSE study, in which our group participated, recently demonstrated the feasibility of two oxygenation strategies in intensive care unit (ICU) patients with ARDS. We have also initiated the LOCO-2 study (NCT02713451), whose aim is to show a reduction in mortality in ARDS using a "conservative" oxygenation strategy (PaO2 maintained between 55 and 70 mmHg) as compared to a classical "liberal" oxygenation strategy (PaO2 between 90 and 105 mmHg).

The LTO-BLOXY study is a substudy of the on-going LOCO-2 study

DETAILED DESCRIPTION:
The LTO-BLOXY study will compare respiratory, cognitive and exercise function outcomes in patients who underwent one of the two oxygenation strategies in the context of the on-going LOCO-2 study:

* Experimental group: oxygenation will be maintained at a level between 55 and 70 mmHg of PaO2 as measured by blood gas test ("conservative" oxygenation). Between blood gas measures, oxygenation will be optimized to achieve an SpO2 between 88% and 92%.
* Control group: oxygenation will be maintained at a level between 90 and 105 mmHg of PaO2 as measured by blood gas test ("liberal" oxygenation). Between blood gas measures, oxygenation will be optimized to achieve an SpO2 >96%.

The primary objective is to demonstrate a lower level of impairment of respiratory function at 6 months in survivors of acute respiratory distress syndrome (ARDS) after a "conservative" oxygenation strategy, as compared to a "liberal" oxygenation strategy.

Secondary objectives are numerous and will explore different areas such as evalution of disability, respiratory function, exercise function, cognitive function and quality of life.

Participation in the LTO-BLOXY study will be proposed to all patients included in LOCO-2 at discharge from the ICU. A total of 259 patients from the overall total of 850 expected inclusions in LOCO-2, will participate in the LTO-BLOXY study. These patients will be followed up to 1 year after their initial inclusion in LOCO-2, with a view to evaluate respiratory function, exercise function and cognitive function, as well as QoL.

The calendar of their study participation is as follows:

* Inclusion in LOCO-2 study and randomization LOCO-2
* Inclusion in LTO-BLOXY study at discharge from the ICU
* 3 month visit ± 2 weeks (3 months after inclusion in LOCO-2 study)
* 6 month visit ± 2 weeks (6 months after inclusion in LOCO-2 study)
* 12 month visit ± 2 weeks (12 months after inclusion in LOCO-2 study)

At each follow-up visit, the patient will attend a consultation in the Department of Physiology - Functional Explorations, where the study questionnaires will be given to the patient for completion. The neuropsychologist will perform the cognitive tests, the respiratory function and exercise tests will also be performed at the same visit.

ELIGIBILITY:
Inclusion Criteria:

* ARDS defined as a PF ratio <300
* Patients under ventilation for <12 hours
* Stabilization period of 3 hours with standardization of ventilation parameters

Inclusion criterion specific for neurological evaluation:

- Patient aged between 20 and 89 years

Exclusion Criteria:

* Chronic respiratory failure or on home ventilation (excluding obstructive sleep apnoea)
* Cardiac arrest
* Moribund patients (death likely within 48 hours as assessed by the ICU physician)
* Gaseous embolism
* CO poisoning
* Pregnant women
* Indication for hyperbaric oxygen treatment
* Persistent pneumothorax
* Gaseous gangrene
* DNR or limited care order

Exclusion criteria specific for neurological evaluation:

* History of neurological disorders: cranial trauma, stroke, cerebral tumor, epilepsy, neuro-degenerative disease.
* Psychiatric disorders: bipolar disorder, psychosis, addiction, schizophrenia.
* Lack of autonomy due to previously documented cognitive and/or psychomotor impairment.
* Hearing and/or sight impairment that prevent the patient from performing the study tests

Patients presenting exclusion criteria for the neurological evaluation can nonetheless be included in the study for the evaluation of respiratory function.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 259 (Estimated)
Dates: Start 2017-09-20 (Actual); Primary Completion 2021-03-20 (Estimated); Study Completion 2021-09-20 (Estimated)

PRIMARY OUTCOMES:
Diffusing Capacity of the Lungs for carbon monoxide (DLCO) | 6 months
  The primary endpoint is the diffusing capacity of the lungs for carbon monoxide (DLCO), a measure that reflects disorders in pulmonary gas volume, the alveolar-capillary membrane, and the volume of blood in the lung capillaries

SECONDARY OUTCOMES:
Evaluation of disability (Functional Independence Measure) | inclusion, 6 months
  FIM scale to assess the patient's performance in the activities of daily living, including cognitive and relational aspects.
A binary composite morbi-mortality variable | 6 months, 12 months
  A binary composite morbi-mortality variable defined as follow:
  * Failure: death or poor FIM
  * Success: alive and good recuperation
Respiratory function: plethysmography | 3 months, 6 months, 12 months
  Total lung capacity and functional residual capacity measured by plethysmography
Respiratory function | 3 months, 6 months, 12 months
  FEV1 and FEV1/FVC ratio
Respiratory function: blood gases | 3 months, 6 months, 12 months
  PaO2 and PaCO2 measured in room air at rest
Respiratory function: inspiratory pressure | 3 months, 6 months, 12 months
  Sniff nasal inspiratory pressure (SNIP) and maximal inspiratory pressure (PImax) (diaphragm function).
Exercise function: 6-min walk test | 3 months, 6 months, 12 months
  distance covered during a 6-minute walk test, in meters
Exercise function: cyclo ergometer | 6 months
  Physiological parameters measured at peak effort limited by symptoms on a bicycle ergometer exercise test
Cognitive function: screening tests | inclusion, 3 months
  Cognitive function will be investigated firstly through the use of rapid screening tests
Cognitive function | 12 months
  Cognitive function will be investigated secondly through an evaluation performed by a neuropsychologist through the use of the RAPID battery
Quality of life: The Medical Outcomes Study 36-Item Short-Form Health Survey (SF-36) | 3 months, 6 months, 12 months
  The SF36, in its validated French language version, is an established instrument used to evaluate quality of life (QoL).The questionnaire yields an overall score between 0 and 100, with a higher score indicating better QoL.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Besançon, Besançon, France